CLINICAL TRIAL: NCT03704974
Title: The Impact of Evidence-Based Parent Training on Pediatric Health Services Utilization
Brief Title: The Impact of Parent Training on the Child's Health Services
Status: Terminated | Type: Observational
Why Stopped: Current high clinical demands of PI.
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: AltaMed Health Services Corporation (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Dean Coffey, Principal Investigator, Children's Hospital Los Angeles
Other Study IDs: CHLA-17-00001; UL1TR001855 (NIH)
Record Dates: First submitted 2018-07-02; First posted 2018-10-15 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Parenting; Child Rearing; Child Behavior Problem
Keywords: Child Health Services; Pediatric Health Service Utilization; Incredible Years

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children of Parents Receiving IY: Children ages 3 to 6 years at start of group with behavior concerns whose parents are referred by their pediatricians for participation in a video-based parent training program from 2014 through 2018.
  Interventions: Behavioral: Video-Based Parent Training Program

INTERVENTIONS:
Behavioral: Video-Based Parent Training Program — An18-20 week evidence-based social cognitive theory-based parenting program where parents see brief video vignettes of effective and less effective parenting and develop concepts to modify their child's behavior.
  Other Names: Incredible Years® Preschool BASIC Parenting Program; Incredible Years® Early Childhood BASIC Parenting Program

SUMMARY:
The purpose of the study is to determine whether parent training with the Incredible Years Parent Program delivered in pediatric primary care decreases usage of healthcare services for the next year when compared to annual healthcare service use during the two years prior to the parents participating in program.

DETAILED DESCRIPTION:
Pediatric health services utilization (pHSU) by children with mental health conditions demonstrated dramatic increases between 2006 and 2011. These national trends reflecting large increases in pHSU for mental health conditions were seen across multiple developmental levels. Health services costs for children with mental health conditions are estimated to be twice those for the average child. The Incredible Years® Parent Program (IY) has a strong evidence-base supporting its effectiveness in reducing early onset conduct problems. The overall objective of this stage 3 (T3) translational research proposal is to conduct a pilot study of 45 pediatrician-referred parents who participate in IY and examine the impact of IY on pHSU of their children. Pediatric HSU outcome measures include: all-cause ED visits; in-patient hospitalizations and length of stay; authorizations for specialist referrals; primary and acute care visits; and ED visits for mental health conditions. The investigator's central hypothesis is that children ages 3 to 6 years with behavior concerns whose parents are referred by their pediatricians for participation in IY will have decreased mean annual all-cause pHSU and decreased ED visits for mental health conditions in the 12 months following IY, compared to the 24 months prior to IY participation. This is important to demonstrate because significant financial barriers exist to integrating effective family focused prevention services like IY into pediatric primary care settings. Demonstration of reduced pHSU is one way to address these translational barriers. Results of this pilot study are expected to provide preliminary data on pre- and post-intervention effect sizes; these data will be used to demonstrate the feasibility of collecting data using existing sources of pHSU to design a more fully powered multi-site trial with a robust comparator group.

ELIGIBILITY:
Inclusion Criteria:

* Children receiving primary care at CHLA AltaMed with parent-reported behavioral concerns whose parents are referred by their pediatricians for participation in the Incredible Years Parenting Program.
* Continuous enrollment in AltaMed Medicaid funded health services during the 24 months prior to participation in IY and 12 months following participation in IY with lapses in coverage of no more than 90 days in length.
* Parents are English or Spanish-speaking or willing to use interpretation if they speak another language.

Exclusion Criteria:

* Private (commercial non-Medicaid) insurance coverage for greater than 90 days during the 24 months prior to participation in IY and 12 months following participation in IY.

Ages: 36 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children participating in the study will be referred from the AltaMed Federally Qualified Health Center, which manages the primary pediatric care at Children's Hospital Los Angeles for 20,000 children who generate 85,000 outpatient visits per year. The population reflects the diversity of Los Angeles County and is predominantly Latino.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Change in Annual Pediatric Health Services Utilization from 24 months prior to IY Parent Group Participation to 12 months following IY Parent Group Participation | Utilization for 24 months prior to intervention and 12 months following intervention
  (1) all-cause Emergency Department (ED) visits (yes/no) and number; (2) ED visits for mental health conditions (yes/no) and number; (3) in-patient hospitalizations (yes/no) and number, and length of stay in days; (4) authorizations for specialist referrals from AltaMed (yes/no) and number; (5) number of AltaMed primary care visits; (6) AltaMed acute care visits (yes/no) and number; (7) AltaMed mental health visits (yes/no) and number; (8) Children's Hospital Los Angeles (CHLA) specialty mental health visits (yes/no) and number.

SECONDARY OUTCOMES:
Eyberg Child Behavior Inventory | During week before or after starting group; and during week before or after ending group, up to 20 weeks
  Raw and T-scores for Intensity [measures frequency of problem behaviors; range 36 to 252; higher worse] and Problem [measures number of behaviors that are a problem for the parent; range 0 to 36; higher worse] Subscales
Youth Outcome Questionnaire (Parent Report) | During week before or after starting group; and during week before or after ending group, up to 20 weeks
  Total raw score [measures change in frequency of child symptoms and prosocial behaviors; range -16 to 240; higher worse].
Pediatric Symptom Checklist | During week before or after starting group; and during week before or after ending group, up to 20 weeks
  Total raw score [measures frequency of pediatric psychosocial problems; range 0 to 70; higher worse].

CONTACTS AND LOCATIONS:
Overall Officials: DEAN M COFFEY, PsyD, MS, Principal Investigator — University of Southern California; Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan approved by our Institutional Review Board (IRB) for sharing individual participant data.

REFERENCES:
- [Background] General US. Mental health: A report of the surgeon general. Rockville, MD: US Department of Health and Human Services. Substance Abuse and Mental Health Services Administration, Center for Mental Health Services, National Institutes of Health, National Institute of Mental Health. 1999.
- [Background] US Department of Health and Human Services. The national survey of children's health 2007. US Department of Health and Human Services, Health Resources and Service Administration, Maternal and Child Health Bureau, Rockville, MD. 2009.
- [Background] Saxena S, Thornicroft G, Knapp M, Whiteford H. Resources for mental health: scarcity, inequity, and inefficiency. Lancet. 2007 Sep 8;370(9590):878-89. doi: 10.1016/S0140-6736(07)61239-2. PMID 17804062
- [Background] Perou R, Bitsko RH, Blumberg SJ, Pastor P, Ghandour RM, Gfroerer JC, Hedden SL, Crosby AE, Visser SN, Schieve LA, Parks SE, Hall JE, Brody D, Simile CM, Thompson WW, Baio J, Avenevoli S, Kogan MD, Huang LN; Centers for Disease Control and Prevention (CDC). Mental health surveillance among children--United States, 2005-2011. MMWR Suppl. 2013 May 17;62(2):1-35. PMID 23677130
- [Background] Torio CM, Encinosa W, Berdahl T, McCormick MC, Simpson LA. Annual report on health care for children and youth in the United States: national estimates of cost, utilization and expenditures for children with mental health conditions. Acad Pediatr. 2015 Jan-Feb;15(1):19-35. doi: 10.1016/j.acap.2014.07.007. Epub 2014 Nov 13. PMID 25444653
- [Background] Fox SE, Levitt P, Nelson CA 3rd. How the timing and quality of early experiences influence the development of brain architecture. Child Dev. 2010 Jan-Feb;81(1):28-40. doi: 10.1111/j.1467-8624.2009.01380.x. PMID 20331653
- [Background] Hertzman C, Boyce T. How experience gets under the skin to create gradients in developmental health. Annu Rev Public Health. 2010;31:329-47 3p following 347. doi: 10.1146/annurev.publhealth.012809.103538. PMID 20070189
- [Background] Yousafzai AK, Rasheed MA, Rizvi A, Armstrong R, Bhutta ZA. Effect of integrated responsive stimulation and nutrition interventions in the Lady Health Worker programme in Pakistan on child development, growth, and health outcomes: a cluster-randomised factorial effectiveness trial. Lancet. 2014 Oct 4;384(9950):1282-93. doi: 10.1016/S0140-6736(14)60455-4. Epub 2014 Jun 16. PMID 24947106
- [Background] Webster-Stratton, C. The Incredible Years®: parents, teachers and children training series. Leader's guide: Preschool version of BASIC. 2008. Seattle, WA
- [Background] Reid MJ, Webster-Stratton C, Baydar N. Halting the development of conduct problems in head start children: the effects of parent training. J Clin Child Adolesc Psychol. 2004 Jun;33(2):279-91. doi: 10.1207/s15374424jccp3302_10. PMID 15136193
- [Background] Reid MJ, Webster-Stratton C, Beauchaine TP. Parent training in head start: a comparison of program response among African American, Asian American, Caucasian, and Hispanic mothers. Prev Sci. 2001 Dec;2(4):209-27. doi: 10.1023/a:1013618309070. PMID 11833925
- [Background] Scott S, Briskman J, O'Connor TG. Early prevention of antisocial personality: long-term follow-up of two randomized controlled trials comparing indicated and selective approaches. Am J Psychiatry. 2014 Jun;171(6):649-57. doi: 10.1176/appi.ajp.2014.13050697. PMID 24626738
- [Background] Scott S, Spender Q, Doolan M, Jacobs B, Aspland H. Multicentre controlled trial of parenting groups for childhood antisocial behaviour in clinical practice. BMJ. 2001 Jul 28;323(7306):194-8. doi: 10.1136/bmj.323.7306.194. PMID 11473908
- [Background] Scott S, Sylva K, Doolan M, Price J, Jacobs B, Crook C, Landau S. Randomised controlled trial of parent groups for child antisocial behaviour targeting multiple risk factors: the SPOKES project. J Child Psychol Psychiatry. 2010 Jan;51(1):48-57. doi: 10.1111/j.1469-7610.2009.02127.x. Epub 2009 Sep 1. PMID 19732250
- [Background] Webster-Stratton C. Preventing conduct problems in Head Start children: strengthening parenting competencies. J Consult Clin Psychol. 1998 Oct;66(5):715-30. doi: 10.1037//0022-006x.66.5.715. PMID 9803690
- [Background] Webster-Stratton C, Rinaldi J, Jamila MR. Long-Term Outcomes of Incredible Years Parenting Program: Predictors of Adolescent Adjustment. Child Adolesc Ment Health. 2011 Feb;16(1):38-46. doi: 10.1111/j.1475-3588.2010.00576.x. PMID 21499534
- [Background] Soni A. The Five Most Costly Children's Conditions, 2011: Estimates for U.S. Civilian Noninstitutionalized Children, Ages 0-17. 2014 Apr. In: Statistical Brief (Medical Expenditure Panel Survey (US)) [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2001-. STATISTICAL BRIEF #434. Available from http://www.ncbi.nlm.nih.gov/books/NBK476257/ PMID 29360325
- [Background] Kubicek K, Liu D, Beaudin C, Supan J, Weiss G, Lu Y, Kipke MD. A profile of nonurgent emergency department use in an urban pediatric hospital. Pediatr Emerg Care. 2012 Oct;28(10):977-84. doi: 10.1097/PEC.0b013e31826c9aab. PMID 23023463
- [Background] Webster-Stratton C, Reid MJ, Beauchaine TP. One-year follow-up of combined parent and child intervention for young children with ADHD. J Clin Child Adolesc Psychol. 2013;42(2):251-61. doi: 10.1080/15374416.2012.723263. Epub 2012 Sep 28. PMID 23020199
- [Background] McCart MR, Priester PE, Davies WH, Azen R. Differential effectiveness of behavioral parent-training and cognitive-behavioral therapy for antisocial youth: a meta-analysis. J Abnorm Child Psychol. 2006 Aug;34(4):527-43. doi: 10.1007/s10802-006-9031-1. Epub 2006 Jul 13. PMID 16838122
- [Background] Menting AT, Orobio de Castro B, Matthys W. Effectiveness of the Incredible Years parent training to modify disruptive and prosocial child behavior: a meta-analytic review. Clin Psychol Rev. 2013 Dec;33(8):901-13. doi: 10.1016/j.cpr.2013.07.006. Epub 2013 Jul 22. PMID 23994367
- [Background] American Academy of Child and Adolescent Psychiatry Committee on Health Care Access and Economics Task Force on Mental Health. Improving mental health services in primary care: reducing administrative and financial barriers to access and collaboration. Pediatrics. 2009 Apr;123(4):1248-51. doi: 10.1542/peds.2009-0048. No abstract available. PMID 19336386
- [Background] Leslie LK, Mehus CJ, Hawkins JD, Boat T, McCabe MA, Barkin S, Perrin EC, Metzler CW, Prado G, Tait VF, Brown R, Beardslee W. Primary Health Care: Potential Home for Family-Focused Preventive Interventions. Am J Prev Med. 2016 Oct;51(4 Suppl 2):S106-18. doi: 10.1016/j.amepre.2016.05.014. Epub 2016 Aug 3. PMID 27498167
- [Background] Case A, Fertig A, Paxson C. The lasting impact of childhood health and circumstance. J Health Econ. 2005 Mar;24(2):365-89. doi: 10.1016/j.jhealeco.2004.09.008. Epub 2005 Jan 5. PMID 15721050
- [Background] Patel V, Flisher AJ, Hetrick S, McGorry P. Mental health of young people: a global public-health challenge. Lancet. 2007 Apr 14;369(9569):1302-1313. doi: 10.1016/S0140-6736(07)60368-7. PMID 17434406
- [Background] Dawson G, Ashman SB, Carver LJ. The role of early experience in shaping behavioral and brain development and its implications for social policy. Dev Psychopathol. 2000 Autumn;12(4):695-712. doi: 10.1017/s0954579400004089. PMID 11202040
- [Background] Champagne FA, Weaver IC, Diorio J, Dymov S, Szyf M, Meaney MJ. Maternal care associated with methylation of the estrogen receptor-alpha1b promoter and estrogen receptor-alpha expression in the medial preoptic area of female offspring. Endocrinology. 2006 Jun;147(6):2909-15. doi: 10.1210/en.2005-1119. Epub 2006 Mar 2. PMID 16513834
- [Background] Walker SP, Wachs TD, Grantham-McGregor S, Black MM, Nelson CA, Huffman SL, Baker-Henningham H, Chang SM, Hamadani JD, Lozoff B, Gardner JM, Powell CA, Rahman A, Richter L. Inequality in early childhood: risk and protective factors for early child development. Lancet. 2011 Oct 8;378(9799):1325-38. doi: 10.1016/S0140-6736(11)60555-2. Epub 2011 Sep 22. PMID 21944375
- [Background] Kershaw P, Irwin L, Trafford K, Hertzman C. The British Columbia atlas of child development (Vol. 40). Vancouver, BC: Human Early Learning Partnership; 2005.
- [Background] Eyberg SM, Pincus D. Eyberg child behavior inventory and sutter-eyberg student behavior inventory-revised: Professional manual. Psychological Assessment Resources; 1999.
- [Background] Wells MG, Burlingame GM, Lambert MJ, Hoag MJ, Hope CA. Conceptualization and measurement of patient change during psychotherapy: Development of the Outcome Questionnaire and Youth Outcome Questionnaire. Psychotherapy: Theory, Research, Practice, Training. 1996;33(2):275. doi:10.1037/0033-3204.33.2.275
- [Background] Jellinek MS, Murphy JM, Little M, Pagano ME, Comer DM, Kelleher KJ. Use of the Pediatric Symptom Checklist to screen for psychosocial problems in pediatric primary care: a national feasibility study. Arch Pediatr Adolesc Med. 1999 Mar;153(3):254-60. doi: 10.1001/archpedi.153.3.254. PMID 10086402
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- See also: Link to REDCap Database — https://redcap.sc-ctsi.org/